CLINICAL TRIAL: NCT05918302
Title: Efficacy, Safety and Patient-reported Outcomes of Peptide Receptor Radionuclide Therapy With 177Lu-edotreotide Compared to Everolimus in Somatostatin Receptor Positive Neuroendocrine Tumors of the Lung and Thymus.
Brief Title: Efficacy and Safety of Radiotherapy Compared to Everolimus in Somatostatin Receptor Positive Neuroendocrine Tumors of the Lung and Thymus.
Acronym: LEVEL
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Grupo Espanol de Tumores Neuroendocrinos (Other)
Collaborators: ITM Oncologics GmbH (Industry); MFAR (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GETNE-T2217; 2022-502154-13-00 (Other: EU CT (CTIS))
Record Dates: First submitted 2023-03-06; First posted 2023-06-26 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-09

CONDITIONS: Neuroendocrine Tumors; Lung Neuroendocrine Neoplasm; Thymus Neoplasms
MeSH Terms: conditions — Neuroendocrine Tumors; Thymus Neoplasms | interventions — 177Lu-octreotide, DOTA(0)-Tyr(3)-; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm (Experimental): Treatment with 6 cycles of 7.5 ± 0.7 GBq 177Lu-edotreotide. The prescribed treatment administration is as follows: a 6 (±2) weeks interval between cycles 1 and 2 followed by all remaining cycles (3-6) given 8 (± 1) weeks after the previous cycle), where possible, or until disease progression, intolerable toxicity or death, whichever occurs first.
  Interventions: Drug: 177Lu-edotreotide
- Control arm (Active Comparator): Everolimus 10 mg orally once daily (QD) until disease progression or intolerable toxicity or death, whichever occurs first.
  Interventions: Drug: Everolimus

INTERVENTIONS:
Drug: 177Lu-edotreotide — 6 cycles of 7.5 ± 0.7 Giga becquerel (GBq) 177Lu-edotreotide
  Arms: Experimental arm
Drug: Everolimus — 10 mg orally once daily (QD)
  Arms: Control arm

SUMMARY:
LEVEL trial aims to demonstrate the higher efficacy of 177Lu-edotreotide over everolimus in patients with well to moderately differentiated neuroendocrine tumors of the lung and thymus who require systemic therapy. It is hypothesized that 177Lu-edotreotide may significantly increase the progression-free survival (PFS) compared to everolimus in lung and thymic carcinoids.

DETAILED DESCRIPTION:
The LEVEL Trial is a randomized, prospective, international, open-label, phase III study comparing everolimus and 177Lu-edotreotide in advanced somatostatin receptor positive (SSTR+) lung and thymic well differentiated neuroendocrine tumors with high expression of somatostatin receptors confirmed by positron emission tomography somatostatin receptor imaging.

In the investigator's opinion, patients recruited into the trial must be eligible to receive everolimus. Patients with both functional and nonfunctional lung and thymus neuroendocrine tumors (NETs) will be included in this trial. In total, 120 patients will be randomized in a 3:2 proportion to either experimental or control arms, respectively.

Randomization will be stratified according to prior medical therapy (tumor treatment-naïve [patients who have not received any prior systemic anticancer therapy] versus non-treatment- naïve [patients who have received one or two prior line of systemic anticancer therapy, including somatostatin analogs (SSAs) as anti-tumor treatment]) and histological differentiation (typical versus atypical / well versus moderately differentiated). Stratification according to the functional status is not foreseen considering the poor predictive and prognostic relevance of this criteria on PRRT in the literature.

Diagnosis of progression and tumor burden will be established based on radiological information from morphological imaging (magnetic resonance imaging [MRI] and/or computed tomography [CT]) according to RECIST v1.1. Tumors assessments will be scheduled every 12 ± 2 weeks from randomization (the first scan will be performed after Cycle 2 for the 177Lu-edotreotide until radiologically confirmed progression of the disease, initiation of new subsequent anticancer therapy, or death (whichever comes first). The scanning modality and protocol should be consistent with the baseline scan. Diagnosis of RECIST v1.1 progression will be made by the local investigator. The confirmatory scans should be performed preferably at the next scheduled imaging visit and no less than 4 weeks after the prior assessment of progression (PD) (in the absence of clinically significant deterioration). Additional MRI/CT scans may be performed at any other time if, in the investigator's clinical judgment, PD is suspected. For equivocal findings of progression, treatment may continue until the next scheduled assessment.

In both arms, for a given patient, trial treatment dosing should be discontinued if there is evidence of RECIST v1.1 progression, in case of persistent toxicities or if the patient withdraws consent to continue with treatment. In all cases, if possible, all other protocol scheduled assessments should be continued until the end of the long-term follow-up period, unless the patient explicitly withdraws consent to all trial procedures and follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Institutional Review Board (IRB)/Independent Ethics Committee (IEC) approved written informed consent.
2. Patients ≥ 18 years of age.
3. Patients who have histologically confirmed metastatic or locally advanced unresectable well/moderately differentiated; World Health Organization (WHO]) 2015 criteria; neuroendocrine tumor of lung (typical and atypical carcinoids) or thymus origin either functioning or non-functioning.
4. Patients must have the appropriate pathological features based on WHO classification, and description of proliferation activity as indicated by mitotic count per 10 high-power fields (HPF) and presence of necrosis, or Ki67 index.
5. In SSTR imaging all RECIST v1.1 selected target lesions and all other lesions considered dominant by the investigator should be positive. If an fluorodeoxyglucose (FDG)-positron emission tomography (FDG-PET) is performed (not mandatory), all FDG-PET positive RECIST v1.1 target lesions and all other FDG-PET positive lesions considered dominant by the investigator should also be positive in SSRT imaging.
6. Lesions must have shown radiological evidence of disease progression in the 12 months prior to inclusion in the study. Patients who were receiving systemic anticancer therapy, progression should be documented on therapy or after stopping therapy due to adverse events or other reasons. Patients without prior therapy, documentation of progression is also mandatory to watch and wait strategy or during the follow up after surgery.
7. Patients may be included in first-line therapy (systemic treatment naïve) or may have experienced progression on somatostatin analogues or additional systemic treatments, which may include but not limited to chemotherapy, targeted agents or immunotherapy (maximum of 2 prior systemic anti-tumor treatments).

   Note: Somatostatin analogues for patients with functioning tumors are allowed.
8. Patients have radiographically documented and measurable metastatic or locally advanced disease at baseline according to RECIST v1.1.
9. An archival tumor tissue sample should be available for submission to the central laboratory prior to study treatment (36 months). If an archival tumor tissue sample is not available, a new biopsy tissue sample should be provided if feasible.
10. Patients who have Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
11. Adequate organ and bone marrow function based upon meeting all of the following laboratory criteria:

    1. Neutrophil count (ANC) ≥ 1,500/mm^3
    2. Platelet count ≥ 75 × 10^9/L
    3. Hemoglobin ≥ 8 g/dL
    4. Serum bilirubin ≤ 1.5 × upper limit of normal (ULN) or ≤ 3 × ULN for subjects with Gilbert's disease or liver metastases
    5. Creatinine clearance (CrCl) ≥ 40 mL/min as estimated by the Cockcroft-Gault formula or as measured by 24-hour urine collection (GFR can also be used instead of CrCl). Note: renal tract obstruction is not allowed.
    6. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN or ≤ 5 x ULN for subjects with liver metastases
12. Female subject must provide a negative urine pregnancy test at screening, and must agree to use a medically accepted and highly effective birth control method (i.e. those with a failure rate less than 1%) for the duration of the study treatment and for 6 months after the final dose of study treatment.
13. Female patients must agree not to breastfeed or donate ovules starting at screening and throughout the study period, and for at least 6 months after the final study drug administration.
14. Male patients must agree not to donate sperm starting at screening and throughout the study period, and for at least 6 months after the final study drug administration.
15. Male patients with a pregnant or breastfeeding partner(s) must agree to abstinence or use a condom for the duration of the pregnancy or time the partner is breastfeeding throughout the study period and for at least 6 months after the final study drug administration.
16. Subject agrees not to participate in another interventional study while on treatment in the present study.

Exclusion Criteria:

1. Patients who are not able to swallow tablets.
2. Patients with poorly-differentiated or high-grade neuroendocrine carcinoma (i.e. large cell neuroendocrine carcinoma of lung, small cell lung cancer) or mixed tumors (i.e. adenocarcinoid tumor) are not eligible.
3. Patients with brain mets unless stable on treatment for > 12 weeks and with no evidence of raised intracranial pressure or mass effect.
4. Patients who have ongoing clinically significant toxicity (Grade 2 or higher with the exception of alopecia) associated with prior treatment (including systemic therapy, radiotherapy or surgery).
5. Patients who have a recent diagnosis of another malignancy (within 12 months prior to inclusion), patients who are on active treatment for other cancer before the first dose of study drug, or any evidence of residual disease from a previously diagnosed malignancy.
6. Patients who have a known active Hepatitis B (e.g., HBsAg reactive) or active hepatitis C (e.g., hepatitis C virus (HCV) RNA [qualitative] is detected). Patients who have a known history of human immunodeficiency virus (HIV) infection (HIV 1 or 2).
7. Patients who have received a live vaccine up to 4 weeks prior to the first dose of trial treatment.

   Note:Live attenuated vaccines should not be administered during the trial treatment and over the next 3 months after the last treatment dose.
8. Patients who have documented history of a cerebral vascular event (stroke or transient ischemic attack), unstable angina, myocardial infarction, or cardiac symptoms (including congestive heart failure) consistent with New York Heart Association Class III-IV within 6 months prior to the first dose of study drug.
9. Prior peptide receptor radionuclide therapy (PRRT) or mammalian target of rapamycin (mTOR) inhibitors (e.g. deforolimus, everolimus, sirolimus, temsirolimus, etc.); or hepatic radio-embolization (within 6 months prior to first dose of study treatment).
10. Prior radiotherapy or major surgery within 12 weeks prior to the first dose of study drug.
11. Patients who have had chemotherapy, biologics, investigational agents, and/or antitumor treatment with immunotherapy that is not completed 4 weeks prior to the first dose of study drug.
12. Patients who have known hypersensitivity to Everolimus or to any excipient contained in the drug formulation of Everolimus.
13. Patients who have known hypersensitivity to 177Lu-edotreotide or to any excipient contained in the drug formulation of 177Lu-edotreotide or the nephroprotective amino acid solution (AAS).
14. Current spontaneous urinary incontinence preventing safe administration of the investigational medicinal product (IMP), in the investigator's opinion.
15. Patients who have other underlying medical conditions that, in the opinion of the investigator, would impair the ability of the subject to receive or tolerate the planned treatment and follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-10-27 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Throughout the study period, approximately 3 years per patient
  Progression-free survival (PFS) defined as the time from the date of randomization to the date of first documentation of disease progression according to RECIST 1.1 by investigator-assessment or death due to any cause, whichever occurs first. In the primary analysis, PFS will be censored at the date of the last adequate tumor assessment if no PFS event is observed prior to the analysis cut-off date.

SECONDARY OUTCOMES:
Objective response rate (ORR) | Throughout the study period, approximately 3 years per patient
  Assessed by the investigator through imaging follow-up (CT scan/MRI) using RECIST v1.1. This will be considered as the percentage/proportion of randomized patients with confirmed complete response (CR) or partial response (PR) as their overall best response throughout the study period.
Disease control rate (DCR) | Throughout the study period, approximately 3 years per patient
  Percentage/proportion of randomized patients with complete response (CR) or partial response (PR), according to ORR definition for the trial, or maintained stable disease (SD) as their overall best response, assessed by imaging follow-up (CT scan/MRI) and RECIST v1.1 criteria. Stable disease should be maintained for at least 4 months to be considered as a DCR event.
Duration of response (DoR) | Throughout the study period, approximately 3 years per patient
  Time from first confirmed response (CR or PR), according to ORR definition for the trial, to the date of the documented PD as determined using RECIST v1.1 criteria or death due to any cause, whichever occurs first. Those patients with response and without PD or death event will be censored on the date of their last tumor assessment.
Overall Survival (OS) | Throughout the study period, approximately 3 years per patient, at each visit. Long-term follow-up to be performed at least every 6 months.
  Defined as the time elapsed from randomization until death from any cause. We will assess the median OS, estimated by Kaplan-Meier. Patients alive and free of events at the date of the analysis will be censored at their last known contact.
Patient reported quality of life | Throughout the study period, approximately 3 years per patient. Assessed every 12 weeks from randomization to progression
  Assessed through the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (QLQ) C30 (EORTC QLQ-C30), version 3 and lung cancer specific extension module LC-13. This are structural questionnaires self completed by the patient and which will give a numerical value to their own perception of quality of life. The scores obtained are standardized and a score between 0 (worst quality of life) and 100 (better quality of life).

CONTACTS AND LOCATIONS:
Overall Officials: Jaume Capdevila, M.D. Ph.D., Study Chair — Hospital Vall d'Hebron
Locations (25):
- Belgium (2):
  - Antwerp University Hospital (UZA), Edegem, Edegem
  - CHU Liège, Liège
- France (8):
  - Hospital Center University Dijon Bourgogne (CHU Bourgogne), Dijon, Dijon
  - Centre Hospitalier Universitaire (CHU) Bordeux, Bourdeaux
  - Lille University Hospital, Lille
  - Hôpital Edouard Herriot, Lyon, Lyon
  - Department of Nuclear Medicine, La Timone University Hospital, CERIMED, Aix-Marseille University, France, Marseille
  - Department of Digestive Oncology, CHU Saint Eloi, Montpellier, France/ ICM Cancer Institute at Montpellier, Montpellier
  - Centre Hospitalier Universitaire de Nantes, Nantes
  - I. Gustave Roussy, Paris, Paris
- Italy (5):
  - Azienda USL IRCCS Di Reggio Emilia, Reggio Emilia, Reggio Emilia
  - IRCCS Istituto Romagnolo per lo Studio dei Tumori "Dino Amadori" - Irsì - Meldola, Meldola
  - Istituto Europeo di Oncologia - Milano, Milan
  - Digestive Disease Unit, Sant'Andrea University Hospital, ENETS Center of Excellence Rome, Rome, Italy., Roma
  - Azienda Ospedaliera Universitaria Integrata Verona, Verona
- Spain (10):
  - Hospital Universitario Virgen del Rocío, Seville, Andalusia
  - ICO Institut Català d'Oncologia L'Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - Complexo Hospitalario Universitario de Santiago de Compostela, Santiago de Compostela, Galicia
  - Hospital General Universitario Gregorio Marañón, Madrid, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid, Madrid, Madrid
  - Fundación Jiménez Díaz University Hospital, Madrid, Madrid
  - Hospital Universitario 12 de Octubre, Madrid, Madrid
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Universitario y Politécnico La Fe, Valencia, Valencia
  - Hospital Universitari Vall d'Hebron, Barcelona

IPD SHARING:
Plan to Share IPD: No
Analyzed compiled results will be publicly available to support the conclusion from the study.
  Individual data will be available upon reasonable request.

REFERENCES:
- [Derived] Capdevila J, Pubul V, Anido U, Walter T, Molina-Cerrillo J, Alonso-Gordoa T, Garcia-Carbonero R, San-Roman-Gil M, Llana B, Jimenez-Fonseca P, Benavent Vinuales M, Ansquer C, Baudin E, Lepage C, Del Olmo-Garcia M, Ruffinelli JC, Beron A, Haissaguerre M, Deshayes E, Taieb D, Baldari S, Sansovini M, Cingarlini S, Filice A, Panzuto F, Alvarez-Alvarez R, Lousberg L, Aboubakar Nana F, Hernando J, Garcia-Alvarez A, Garcia-Burillo A, Villacampa G, Vandamme T, Fazio N, Durand A. A Randomized clinical trial evaluating the impact on survival and quality of life of 177Lutetium[Lu]-edotreotide versus everolimus in patients with neuroendocrine tumors of the lung and thymus: the LEVEL study (GETNE T-2217). BMC Cancer. 2025 Apr 4;25(1):613. doi: 10.1186/s12885-025-13941-3. PMID 40186126